CLINICAL TRIAL: NCT07047339
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Probiotic 6600 as an Adjuvant Therapy for Colitis
Brief Title: Evaluate the Efficacy and Safety of Probiotic 6600 as an Adjuvant Therapy for Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6600
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colitis; IBD (Inflammatory Bowel Disease); Probiotic Intervention
MeSH Terms: conditions — Colitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- UC control group (Placebo Comparator): Patients diagnosed with ulcerative colitis (UC) were given one tablet of placebo twice daily (morning and evening after meals) with warm water.
  Interventions: Drug: Placebo
- UC experimental group (Experimental): Patients diagnosed with ulcerative colitis (UC) were given probiotics 6600 orally twice daily (morning and evening after meals), one tablet each time, with warm water.
  Interventions: Drug: Probiotics 6600
- CD control group (Placebo Comparator): Patients diagnosed with Crohn's disease (CD) were given one tablet of placebo twice daily (morning and evening after meals) with warm water.
  Interventions: Drug: Placebo
- CD experimental group (Experimental): Patients diagnosed with Crohn's disease (CD) were given probiotics 6600 orally twice a day (morning and evening after meals), one tablet each time, with warm water.
  Interventions: Drug: Probiotics 6600
- Colitis control group (Placebo Comparator): Patients diagnosed with colitis (non-ulcerative colitis or Crohn's disease) were given one tablet of placebo twice daily (morning and evening after meals) with warm water.
  Interventions: Drug: Placebo
- Colitis experimental group (Experimental): For patients diagnosed with colitis (non-ulcerative colitis or Crohn's disease), take probiotic 6600 orally twice daily (morning and evening after meals), one tablet each time, with warm water.
  Interventions: Drug: Probiotics 6600

INTERVENTIONS:
Drug: Probiotics 6600 — As the core commensal bacteria of human body, probiotic 6600 has a unique ability to synthesize adhesins and exopolysaccharides. The intestinal protective effect is mediated by the following mechanisms: (1) regulation of Treg/Th17 balance by producing short-chain fatty acids (SCFAs); (2) activation of TLR2/MyD88 pathway inhibits NF-κB inflammatory cascade; (3) Upregulation of zonula occludens-1 enhances intestinal barrier function. Notably, this strain specifically metabolized arabinoxylan to produce the anti-inflammatory metabolite indole lactate, which has important therapeutic value in the colitis microenvironment.
  Probiotic 6600 capsules are enteric capsules (containing probiotic 6600 10^11 CFU/ capsule), taken orally twice a day (after meals in the morning and evening), one capsule each time, and taken with warm water. The drug was stored at 2-8℃.
  Arms: CD experimental group; Colitis experimental group; UC experimental group
Drug: Placebo — The placebo capsules were also enteric-coated capsules, and were taken orally twice a day (morning and evening after meals), one capsule each time, with warm water.
  Arms: CD control group; Colitis control group; UC control group

SUMMARY:
This study was conducted in two phases. In Phase I, 40 UC participants, 40 CD participants, and 40 colitis participants were randomly assigned in a 1:1 ratio to the experimental group and the control group, respectively. The study included a screening period (1 week), a double-blind treatment period (24 weeks), an exit examination (1 day), and a safety follow-up period (4 weeks). After providing informed consent, participants who met the inclusion criteria and those who did not meet the exclusion criteria were randomly assigned, in a 1:1 ratio, to receive either the trial (probiotic 6600 capsules) or the control group (placebo). The clinical remission rate (SCCAI score ≤2 and no single subscore >1) after 24 weeks of treatment was calculated. Mayo score ≤2 and no single subscore >1; CDAI score ≤2 and no single subscore >1) were used as the primary efficacy index.

ELIGIBILITY:
Inclusion Criteria:

1. Ulcerative colitis (UC) : met the clinical diagnostic criteria of UC "Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (2023, Xi 'an)", and modified Mayo score ≥4 points;
2. Crohn's disease (CD) : met the clinical diagnostic criteria of CD "Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (2023, Guangzhou)", and CDAI score ≥220;
3. Colitis: clinical diagnosis of colitis and modified SCCAI score ≥3; 3.
4. The age of signing the informed consent form was from 18 to 75 years old (including the cut-off value, male and female were not limited);
5. Complete medical history;
6. From the time of informed consent until 3 months after the last dose of dose, the participant committed to not having any plans to have children or to have any plans to donate sperm or eggs, and to voluntarily use non-pharmacologic contraception;
7. Fully understand the content, process and possible adverse reactions of the trial, voluntarily participate in the trial, and sign the informed consent.

Exclusion Criteria:

1. Taking prebiotics or probiotics in the past 2 weeks or allergic to intervention preparations;
2. Short bowel syndrome, abdominal abscess, toxic megacolon, intestinal perforation, active fistula of digestive tract, severe intestinal stenosis with obstructive symptoms, suspected intestinal obstruction, total colectomy;
3. Other autoimmune diseases, hematological diseases, tumors, acute infections, severe hepatic and renal insufficiency (ALT>2 times the upper limit of normal), severe diseases such as neutropenia, heart failure, organic heart disease, viral hepatitis B, liver cirrhosis, renal impairment (serum creatinine > 2mg/dL or 177mmol/L), AIDS And mental disorders;
4. History of psychoactive substance abuse;
5. A history of drug or other dependent substance abuse, or heavy alcohol consumption in the last 2 weeks (i.e. 28 standard units per week for men and 21 standard units per week for women (1 standard unit contains 14g of alcohol, such as 360mL of beer or 25mL of 40% spirits or 150mL of wine); Heavy drinkers during the trial;
6. Pregnant or breastfeeding women, or planning to become pregnant in the next 6 months;
7. Nervous system diseases such as Alzheimer's disease, stroke, Parkinson's disease;
8. Participated in other clinical trials within the past 6 months;
9. Incomplete medical record information (including gender, age, diagnostic information, colonoscopy results, pathological diagnosis results and other demographic data, etc.);
10. Other investigators deemed ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | To evaluate the effect of taking probiotic 6600 capsules in addition to usual care for 24 weeks on improving the rate of clinical remission compared with the control group.
  To evaluate the efficacy of probiotic 6600 capsule in the adjuvant treatment of patients with colitis.
  We assessed the rate of clinical remission (UC group: Mayo score ≤2 and no single subscore >1; CD group: CDAI score < 150; Colitis group: SCCAI score ≤2 and no single subscore >1).

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided